CLINICAL TRIAL: NCT02545127
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Trial Exploring the Efficacy and Safety of Intra-nasal Administration of Merotocin in Increasing Milk Production in Maternal Subjects With Preterm Delivery and Inadequate Milk Production
Brief Title: Merotocin in Mothers With Inadequate Milk Production and Infants Delivered Prematurely
Acronym: MERMAID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely terminated. Termination was not because of safety concerns but due to slow recruitment.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000050
Record Dates: First submitted 2015-08-26; First posted 2015-09-09 (Estimated); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-11

CONDITIONS: Preterm Delivery; Inadequate Milk Production
Keywords: Inadequate Milk Production
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Merotocin (a selective oxytocin-receptor agonist) (Experimental)
  Interventions: Drug: Merotocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Merotocin — Merotocin nasal spray 400 μg/dose, 2 sprays with 1 spray in each nostril administered 6 to 8 times/day (Day 1 to Day 14).
  Other Names: FE 202767
  Arms: Merotocin (a selective oxytocin-receptor agonist)
Drug: Placebo — Placebo nasal spray, 2 sprays with 1 spray in each nostril administered 6 to 8 times/day (Day 1 to Day 14).
  Arms: Placebo

SUMMARY:
Induction and support of lactation in women with preterm delivery and inadequate milk production.

ELIGIBILITY:
Inclusion Criteria:

* Delivered at the hospital system associated with the trial center
* Delivered preterm singleton gestational age 24 weeks + 0 days to 34 weeks + 2 days
* Willing to express milk at least 5 times every 24 hours during the observation period and 6 to 8 times every 24 hours during the treatment and post-treatment follow up
* Produced < 200 mL milk in 24 hours prior to randomization
* Delivered 96 to 192 (+4) hours prior to randomization

Exclusion Criteria:

* Pre-pregnancy body mass index (BMI) > 50 kg/m^2
* Mastitis
* History of breast trauma, breast surgery, nipple piercing
* Prolactin-releasing pituitary tumor, history of Sheehan's syndrome, pituitary surgery/radiation therapy
* Pre-pregnancy insulin-dependent diabetes mellitus, polycystic ovarian syndrome. Note: gestational diabetes is allowed (also when requiring the use of insulin for treatment)
* Unstable thyroid disease
* Moderate or severe renal or hepatic impairment
* Mental illness
* Significant nasal congestion or mucous production
* Use of anti-psychotic drugs within past 12 months

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (10):
- United States (10):
  - Ferring Investigational Site, New Haven, Connecticut
  - Ferring Investigational Site, South Bend, Indiana
  - Ferring Investigational Site, Baltimore, Maryland
  - Ferring Investigational Site, Boston, Massachusetts
  - Ferring Investigational Site, Valhalla, New York
  - Ferring Investigational Site, Raleigh, North Carolina
  - Ferring Investigational Site, Cincinnati, Ohio
  - Ferring Investigational Site, Charleston, South Carolina
  - Ferring Investigational Site, Houston, Texas
  - Ferring Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 12 investigational sites in the US between May 2021 and November 2022.
Pre-assignment Details: In total, 15 participants were screened. Of these, 11 were screening failures and 4 participants were randomized. All the randomized participants were exposed to the investigational medicinal product (IMP): 2 participants to Merotocin and 2 participants to Placebo.
Period: Overall Study
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (1.4) | 31.5 (6.4) | 31.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (2.2) | 31.7 (0.1) | 29.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Volume of Mother's Own Milk (MoM)
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Daily days 1 to 14
Population: The trial was prematurely terminated due to slow recruitment. Data (if collected) are not presented in order to protect the privacy of the trial participant(s).
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to First Occurrence of Daily Volume of MoM ≥ 500 mL
Description: Number of days
Time Frame: From randomization (Day 1) to Day 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to First Occurrence of Daily Volume of MoM ≥ 750 mL
Description: Number of days
Time Frame: From randomization (Day 1) to Day 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Participants With a Daily Volume of MoM ≥ 500 mL
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Days 1 to 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of Participants With a Daily Volume of MoM ≥ 750 mL
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Days 1 to 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Volume of MoM
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Days 15 to 17
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Volume of MoM Fed to the Infant
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Days 1 to 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Volume of Formula/Donor Milk Fed to the Infant
Description: Measured by weight in grams converted to volume in milliliters (mL)
Time Frame: Days 1 to 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Merotocin Concentration in Milk
Time Frame: Day 3
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Merotocin Concentration in Milk
Time Frame: Day 10
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Infant Body Weight
Time Frame: From baseline (Day 1) to Day 14
Population: as for outcome 1
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Frequency of Adverse Events (AEs) in Maternal Participants
Time Frame: From Screening (0-144 hours of delivery) up to Day 18
Measure: Count of Participants; unit: Participants
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 0 | 1

13. Secondary Outcome: Intensity of AEs in Maternal Participants
Time Frame: From Screening (0-144 hours of delivery) up to Day 18
Measure: Number; unit: Severe Adverse Events
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Severe Adverse Events | 0 | 2

14. Secondary Outcome: Frequency of AEs in Infants
Time Frame: From screening until milk expressed Days 1-14 is consumed/discarded or infant discharged from neonatal intensive care unit (NICU), whichever occurs last.
Measure: Count of Participants; unit: Participants
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 0 | 2

15. Secondary Outcome: Intensity of AEs in Infants
Time Frame: as for outcome 14
Measure: Number; unit: Adverse Events
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Adverse Events
  Mild adverse events | 0 | 2
  Moderate adverse events | 0 | 10
  Severe adverse events | 0 | 3

16. Secondary Outcome: Changes in Routine Safety Laboratory Parameters in Maternal Participants
Time Frame: From screening up to Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

17. Secondary Outcome: Proportion of Maternal Participants With Markedly Abnormal Changes in Laboratory Values
Time Frame: From screening up to Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded from the time of signing ICF through the Day 18/Follow-up visit
Arm/Group | Merotocin (a Selective Oxytocin-receptor Agonist) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merotocin (a Selective Oxytocin-receptor Agonist) (N=2) | Placebo (N=2)
Infections NEC (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merotocin (a Selective Oxytocin-receptor Agonist) (N=2) | Placebo (N=2)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT02545127/Prot_SAP_000.pdf